CLINICAL TRIAL: NCT00999869
Title: The Comparison Study of Intralesional Botulinum Toxin A and Corticosteroid Injection for Alopecia Areata
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Rattapon Thuangtong, Assistance professor, Siriraj Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SirirajH-2
Record Dates: First submitted 2009-10-21; First posted 2009-10-22 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Alopecia Areata
Keywords: Newly diagnosed; Alopecia areata; Botulinum toxin A; Corticosteroid; Intralesional injection
MeSH Terms: conditions — Alopecia Areata | interventions — Botulinum Toxins, Type A; Triamcinolone Acetonide; Triamcinolone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Botulinum toxin A (Experimental): At first visit, patients will be randomized by blocked randomization into 2 sides of scalp. Experimental side will be injected with botulinum toxin A ( Botox) 2 units per 6.05 cm2 of lesion ( Concentration 2 units of Botox per 0.1 ml of normal saline ).
  Interventions: Drug: Botulinum toxin type A
- Triamcinolone acetonide (Active Comparator): At visit0, patients will be injection with triamcinolone acetonide concentration at 10 mg/ml on the comparison side
  Interventions: Drug: Triamcinolone acetonide

INTERVENTIONS:
Drug: Botulinum toxin type A — Using concentration at 2 units per 0.1 of dilution with normal saline Injection in the first visit and follow up at 1 week, 1,2,3 and 4 months after injection
  Other Names: Botox( Allergan Inc.)
  Arms: Botulinum toxin A
Drug: Triamcinolone acetonide — Using concentration at 10 mg/ml and equal amount of botulinum toxin A dilution
  Other Names: Kenacort
  Arms: Triamcinolone acetonide

SUMMARY:
Alopecia areata is one of the most common cause of non-scarring alopecia. The pathogenesis is still unclear, however, it is believed to be an autoimmune disease. This disease is not a life-threatening condition but it has a significant psychological impact to patient's quality of life.

Many triggers have been proposed such as viral infection, stress and neurologic factors. There are many studies show the correlation between disease activities and neurotransmitters level. Substance P and calcitonin gene-related peptide play major role in early stage of disease. These substances cause imbalance of CD4/CD8 lymphocyte in pathologic site and loss of immune privilege of hair follicles.

The conventional treatment of alopecia areata with intralesional corticosteroid injection might treat the end of pathogenesis process.

There is no therapeutic intervention for the origin of disease. Fortunately, botulinum toxin A could be a novel treatment of alopecia areata. The botulinum toxin A demonstrates inhibition release of substance P in many publications.

To sum up, the treatment of alopecia areata with intralesional corticosteroid injection still be a standard treatment, nevertheless, patients have to receive this treatment every month until regrowth of scalp hair. Corticosteroid injection have several side effects, for example, skin atrophy, pigmentary change and hypothalamic-pituitary-adrenal axis suppression. Moreover, injection pain is also affect to psychological aspect .

This study purpose is to evaluate the efficacy of botulinum toxin A for alopecia areata and reduce corticosteroid side effects, as well as, others opportunity cost. There is no prospective, randomized-controlled trial of comparison study between botulinum toxin A injection and corticosteroid injection for alopecia areata, therefore, investigators conduct this study for the greatest benefit to alopecia areata patients and for the future research in disease etiology.

DETAILED DESCRIPTION:
Inclusion criteria

1. Patients must be above 18 years old
2. Newly diagnosed with multiple alopecia areata
3. Patient has lesions on the both side of the scalp.
4. Lesions's diameter varies between 2-6 cms

Exclusion criteria

1. Having active scalp inflammation
2. Allergic to botulinum toxin A or human albumin
3. Receiving any medication that interfere efficacy of botulinum toxin such as macrolides antimicrobial agents or neuromuscular medications
4. Diagnosed with neuromuscular diseases such as Myasthenia gravis
5. Pregnant, breast feeding, plan to pregnant patients

ELIGIBILITY:
Inclusion criteria

* Patients must be above 18 years old
* Newly diagnosed with multiple alopecia areata
* Patient has lesions on the both side of the scalp.
* Lesions's diameter varies between 2-6 cms

Exclusion criteria

* Having active scalp inflammation
* Allergic to botulinum toxin A or human albumin
* Receiving any medication that interfere efficacy of botulinum toxin such as macrolides antimicrobial agents or neuromuscular medications
* Diagnosed with neuromuscular diseases such as Myasthenia gravis
* Pregnant, breast feeding, plan to pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-11; Primary Completion 2012-12 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
The percentage of terminal hair regrowth after intralesional botulinum toxin A injection | 4 months

SECONDARY OUTCOMES:
Possible side effects of intralesional botulinum toxin a injection | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Rattapon Thoungtong, MD., Study Chair — Department of Dermatology, Faculty of medicine Siriraj Hospital, Mahidol University,Thailand; Supenya Varothai, MD., Study Director — Department of Dermatology, Faculty of medicine Siriraj Hospital, Mahidol University,Thailand; Rasthawathana Desomchoke, MD., Principal Investigator — Department of Dermatology, Faculty of medicine Siriraj Hospital, Mahidol University,Thailand; Kumpol Aiempanakit, M.D., Principal Investigator — Department of Dermatology, Faculty of medicine Siriraj Hospital, Mahidol University,Thailand
Locations (2):
- Thailand (2):
  - Siriraj hospital, Bangkok, Bangkok
  - Department of Dermatology, Faculty of medicine Siriraj Hospital, Mahidol University, Bangkok

REFERENCES:
- [Background] Safavi KH, Muller SA, Suman VJ, Moshell AN, Melton LJ 3rd. Incidence of alopecia areata in Olmsted County, Minnesota, 1975 through 1989. Mayo Clin Proc. 1995 Jul;70(7):628-33. doi: 10.4065/70.7.628. PMID 7791384
- [Background] McDonagh AJ, Messenger AG. The pathogenesis of alopecia areata. Dermatol Clin. 1996 Oct;14(4):661-70. doi: 10.1016/s0733-8635(05)70392-2. PMID 9238324
- [Background] Jackow C, Puffer N, Hordinsky M, Nelson J, Tarrand J, Duvic M. Alopecia areata and cytomegalovirus infection in twins: genes versus environment? J Am Acad Dermatol. 1998 Mar;38(3):418-25. doi: 10.1016/s0190-9622(98)70499-2. PMID 9520023
- [Background] Delamere FM, Sladden MM, Dobbins HM, Leonardi-Bee J. Interventions for alopecia areata. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD004413. doi: 10.1002/14651858.CD004413.pub2. PMID 18425901
- [Background] Charuwichitratana S, Wattanakrai P, Tanrattanakorn S. Randomized double-blind placebo-controlled trial in the treatment of alopecia areata with 0.25% desoximetasone cream. Arch Dermatol. 2000 Oct;136(10):1276-7. doi: 10.1001/archderm.136.10.1276. No abstract available. PMID 11030789
- [Background] Kar BR, Handa S, Dogra S, Kumar B. Placebo-controlled oral pulse prednisolone therapy in alopecia areata. J Am Acad Dermatol. 2005 Feb;52(2):287-90. doi: 10.1016/j.jaad.2004.10.873. PMID 15692475
- [Background] Lassus A, Eskelinen A, Johansson E. Treatment of alopecia areata with three different PUVA modalities. Photodermatol. 1984 Jun;1(3):141-4. PMID 6527956
- [Background] Mitchell AJ, Douglass MC. Topical photochemotherapy for alopecia areata. J Am Acad Dermatol. 1985 Apr;12(4):644-9. doi: 10.1016/s0190-9622(85)70088-6. PMID 3989026
- [Background] Tosti A, De Padova MP, Minghetti G, Veronesi S. Therapies versus placebo in the treatment of patchy alopecia areata. J Am Acad Dermatol. 1986 Aug;15(2 Pt 1):209-10. doi: 10.1016/s0190-9622(86)70158-8. PMID 3528241
- [Background] Vestey JP, Savin JA. A trial of 1% minoxidil used topically for severe alopecia areata. Acta Derm Venereol. 1986;66(2):179-80. PMID 2424249
- [Background] Fransway AF, Muller SA. 3 percent topical minoxidil compared with placebo for the treatment of chronic severe alopecia areata. Cutis. 1988 Jun;41(6):431-5. PMID 3292159
- [Background] Price VH. Double-blind, placebo-controlled evaluation of topical minoxidil in extensive alopecia areata. J Am Acad Dermatol. 1987 Mar;16(3 Pt 2):730-6. doi: 10.1016/s0190-9622(87)70095-4. PMID 3549809
- [Background] Fiedler-Weiss VC, Buys CM. Evaluation of anthralin in the treatment of alopecia areata. Arch Dermatol. 1987 Nov;123(11):1491-3. PMID 3314718
- [Background] van der Steen PH, van Baar HM, Happle R, Boezeman JB, Perret CM. Prognostic factors in the treatment of alopecia areata with diphenylcyclopropenone. J Am Acad Dermatol. 1991 Feb;24(2 Pt 1):227-30. doi: 10.1016/0190-9622(91)70032-w. PMID 2007667
- [Background] Gupta AK, Ellis CN, Cooper KD, Nickoloff BJ, Ho VC, Chan LS, Hamilton TA, Tellner DC, Griffiths CE, Voorhees JJ. Oral cyclosporine for the treatment of alopecia areata. A clinical and immunohistochemical analysis. J Am Acad Dermatol. 1990 Feb;22(2 Pt 1):242-50. doi: 10.1016/0190-9622(90)70032-d. PMID 2138175
- [Background] Shapiro J, Lui H, Tron V, Ho V. Systemic cyclosporine and low-dose prednisone in the treatment of chronic severe alopecia areata: a clinical and immunopathologic evaluation. J Am Acad Dermatol. 1997 Jan;36(1):114-7. doi: 10.1016/s0190-9622(97)70342-6. No abstract available. PMID 8996277
- [Background] Bui K, Polisetty S, Gilchrist H, Jackson SM, Frederic J. Successful treatment of alopecia universalis with alefacept: a case report and review of the literature. Cutis. 2008 May;81(5):431-4. PMID 18543595
- [Background] Ettefagh L, Nedorost S, Mirmirani P. Alopecia areata in a patient using infliximab: new insights into the role of tumor necrosis factor on human hair follicles. Arch Dermatol. 2004 Aug;140(8):1012. doi: 10.1001/archderm.140.8.1012-a. No abstract available. PMID 15313825
- [Background] Strober BE, Siu K, Alexis AF, Kim G, Washenik K, Sinha A, Shupack JL. Etanercept does not effectively treat moderate to severe alopecia areata: an open-label study. J Am Acad Dermatol. 2005 Jun;52(6):1082-4. doi: 10.1016/j.jaad.2005.03.039. PMID 15928633
- [Background] Price VH, Hordinsky MK, Olsen EA, Roberts JL, Siegfried EC, Rafal ES, Korman NJ, Altrabulsi B, Leung HM, Garovoy MR, Caro I, Whiting DA. Subcutaneous efalizumab is not effective in the treatment of alopecia areata. J Am Acad Dermatol. 2008 Mar;58(3):395-402. doi: 10.1016/j.jaad.2007.10.645. PMID 18280336
- [Background] Fabre C, Dereure O. Worsening alopecia areata and de novo occurrence of multiple halo nevi in a patient receiving infliximab. Dermatology. 2008;216(2):185-6. doi: 10.1159/000111523. Epub 2008 Jan 23. No abstract available. PMID 18216487
- [Background] Cutrer FM, Pittelkow MR. Cephalalgic alopecia areata: a syndrome of neuralgiform head pain and hair loss responsive to botulinum A toxin injection. Cephalalgia. 2006 Jun;26(6):747-51. doi: 10.1111/j.1468-2982.2006.01098.x. No abstract available. PMID 16686916
- [Background] Paus R, Heinzelmann T, Schultz KD, Furkert J, Fechner K, Czarnetzki BM. Hair growth induction by substance P. Lab Invest. 1994 Jul;71(1):134-40. PMID 7518880
- [Background] Olsen E, Hordinsky M, McDonald-Hull S, Price V, Roberts J, Shapiro J, Stenn K. Alopecia areata investigational assessment guidelines. National Alopecia Areata Foundation. J Am Acad Dermatol. 1999 Feb;40(2 Pt 1):242-6. doi: 10.1016/s0190-9622(99)70195-7. No abstract available. PMID 10025752
- [Background] Hsu TS, Dover JS, Arndt KA. Effect of volume and concentration on the diffusion of botulinum exotoxin A. Arch Dermatol. 2004 Nov;140(11):1351-4. doi: 10.1001/archderm.140.11.1351. PMID 15545544